CLINICAL TRIAL: NCT05091450
Title: Efficacy of a Couple-Based Integrative Body-mind-spirit Group Intervention for Infertile Couples on Improving Dyadic Couple Flourishing and Fertility Quality of Life: A Randomized Controlled Trial
Brief Title: Integrative Body-Mind-Spirit Group Intervention for Infertile Couples
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Dr. Celia Hoi-Yan Chan, Associate Professor, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: EA210488
Record Dates: First submitted 2021-10-09; First posted 2021-10-25 (Actual); Last update posted 2022-11-02 (Actual); Status verified 2022-11

CONDITIONS: Infertility
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Couple-based I-BMS intervention for infertility (Experimental): The I-BMS intervention will be conducted face-to-face and in group format. It comprises four 3-hour sessions within one month. Two registered social workers who are professionally trained on I-BMS intervention model will deliver the intervention.
  Interventions: Behavioral: Couple-based I-BMS intervention for infertility
- Waitlist control (Other): Couples allocated in the waitlist control group will begin the I-BMS intervention (same as the intervention group) after completing the 1-month follow-up assessment.
  Interventions: Behavioral: Couple-based I-BMS intervention for infertility

INTERVENTIONS:
Behavioral: Couple-based I-BMS intervention for infertility — It is based on the previous I-BMS intervention for women undergoing IVF treatment, and aims to improve fertility quality of life and couple flourishing by (1) increasing awareness of the interconnectedness between physical and psychosocial well-being, (2) practicing body-mind-spirit techniques, (3) facilitating personal growth and partner empathy and compassion, and (3) creating the shared meaning of life, family, children. As a strength-focused and meaning-oriented approach, it utilizes experiential and self-reflective exercises to help participants reconstruct the meaning behind their ordeal and rediscover the strengths that keep them going.

SUMMARY:
This is a two-arm, with equal randomization, parallel randomized controlled trial. It compares the efficacy of a couple-based Integrative Body-Mind-Spirit (I-BMS) group intervention to a waitlist control group in improving dyadic couple flourishing and fertility-related quality of life among couples who are diagnosed of infertility in Hong Kong. It also aims to investigate the dyadic associations between infertile husbands' and wives' baseline primary outcomes and changes in primary outcomes following the intervention.

DETAILED DESCRIPTION:
Infertility is a global public health issue, affecting approximately 15% of childbearing-aged couples around the world. It is often a challenging dyadic life experience that generates adverse impacts on the psychosocial well-being of couples at childbearing age. Numerous psychosocial interventions have been developed for infertile women, and their efficacy and effectiveness were supported empirically. This study attempts to address the limitations incurred in existing psychosocial interventions for infertility by: (1) including infertile men and couples who have not sought fertility treatment and (2) incorporating relational outcomes within psychosocial interventions for infertile couples. This is a two-arm, with equal randomization, parallel randomized controlled trial. It compares the efficacy of a couple-based Integrative Body-Mind-Spirit (I-BMS) group intervention to a waitlist control group in improving dyadic couple flourishing and fertility-related quality of life among couples who are diagnosed of infertility in Hong Kong. It also aims to investigate the dyadic associations between infertile husbands' and wives' baseline primary outcomes and changes in primary outcomes following the intervention.

On hundred and seventy-eight infertile couples will be recruited through hospitals, clinics and local communities in Hong Kong. Each prospective couple will complete an online screening survey. Eligible couples will complete the baseline assessment, and then be randomized in a ratio of 1:1 into one of the two arms. Arm 1 is the couple-based I-BMS intervention for infertility, which consists of four 3-hour sessions within one month. Arm 2 is the waitlist control. Randomization will be performed by a computer. All eligible couples will be contacted by a research assistant for a pre-group interview prior to the commencement of the I-BMS intervention. The primary outcomes are changes over the measurement points in dyadic couple flourishing and fertility quality of life. The secondary outcomes include changes over the measurement points in empathy towards partner, partnership, relationship satisfaction, anxiety, depression, infertility-related blame, and resilience. Assessments are administered at baseline, post-intervention, 1-month follow-up, and 5-year follow-up. Structural equation modelling will be employed to examine the efficacy of the couple-based I-BMS intervention based on the intention-to-treat principle, as well as the dyadic association between infertile husbands' and wives' primary outcomes.

Eight hypotheses are generated. First, it is hypothesized that, after controlling for baseline dyadic couple flourishing, couples in the I-BMS intervention group will report significantly higher dyadic couple flourishing than their counterparts in the waitlist control group following the intervention. Second, it is hypothesized that, after controlling for post-intervention dyadic couple flourishing, couples in the I-BMS intervention group will report significantly higher dyadic couple flourishing than their counterparts in the waitlist control group at one-month follow-up. Third, it is hypothesized that, after controlling for baseline dyadic fertility quality of life, couples in the I-BMS intervention group will report significantly higher dyadic fertility quality of life than their counterparts in the waitlist control group following the intervention. Fourth, it is hypothesized that, after controlling for post-intervention dyadic fertility quality of life, couples in the I-BMS intervention group will report significantly higher dyadic fertility quality of life than their counterparts in the waitlist control group at one-month follow-up. Fifth, it is hypothesized that wives' baseline fertility quality of life is predicted by their own and their husbands' baseline couple flourishing. Sixth, it is hypothesized that husbands' baseline fertility quality of life is predicted by their own and their wives' baseline couple flourishing. Seventh, it is hypothesized that wives' post-intervention improvements in fertility quality of life is predicted by their own and their husbands' post-intervention improvements in couple flourishing. Eighth, it is hypothesized that husbands' post-intervention improvements in fertility quality of life is predicted by their own and their wives' post-intervention improvements in couple flourishing.

ELIGIBILITY:
Inclusion Criteria (Couples):

* are in a heterosexual marriage
* are clinically diagnosed of infertility
* are actively trying to conceive
* are able to understand, read and speak Chinese
* age 18 or above
* give consent to participate in this study

Exclusion Criteria (Couples):

* are being exposed to intimate partner violence within the past 12 months (HARK test score >=1)
* have signs of early psychosis within the past 12 months (Screen for Early Psychosis score = 2)
* have suicidal ideation in the past 2 weeks (Beck Depression Inventory II, item 9, score >= 2)
* already have a living child or children

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 356 (Estimated)
Dates: Start 2023-07-01 (Estimated); Primary Completion 2025-04-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Changes over the measurement points in the Couple Flourishing Measure | Baseline, post-intervention: 4 weeks after the intervention initiation, 1-month follow-up, 5-year follow-up
  It has 16 items measuring participants' perceived encouragement towards expanding goals, recognition of partner's strengths, and engagement in meaningful activities with their partner. Scores range from 16 to 112, where a higher score represents a higher level of couple flourishing.
Changes over the measurement points in the Fertility Quality of Life Questionnaire - Core FertiQoL subscale | Baseline, post-intervention: 4 weeks after the intervention initiation, 1-month follow-up, 5-year follow-up
  It has 24 items measuring the consequences of fertility problems on quality of life over four life domains (emotional, mind/body, relational, and social). Subscale scores range from 0 to 100, where a higher score represent a higher level of fertility quality of life.

SECONDARY OUTCOMES:
Changes over the measurement points in the Interpersonal Reactivity Index | Baseline, post-intervention: 4 weeks after the intervention initiation, 1-month follow-up, 5-year follow-up
  It has 13 items measuring participants' tendency to view things from their partner's perspective and to have sympathy and concerns for partner's misfortune. Scores range from 0 to 52, where a higher score represent greater perspective taking and empathic concern.
Changes over the measurement points in the Relationship Flourishing Scale | Baseline, post-intervention: 4 weeks after the intervention initiation, 1-month follow-up, 5-year follow-up
  It has 12 items measuring participants' perception that meaningful connections, shared goals, and supportive activities in their relationship have helped each other grow as individuals and as a couple. Scores range from 12 to 60, where a higher score represents a higher level of relationship flourishing.
Changes over the measurement points in the Brief Version of the Dyadic Adjustment Scale | Baseline, post-intervention: 4 weeks after the intervention initiation, 1-month follow-up, 5-year follow-up
  It has 4 items measuring participants' perceived satisfaction towards their marriage. Scores range from 0 to 20, where a higher score represents greater marital satisfaction.
Changes over the measurement points in the Hospital Anxiety and Depression Scale | Baseline, post-intervention: 4 weeks after the intervention initiation, 1-month follow-up, 5-year follow-up
  It has 14 items measuring participants' levels of anxiety and depression. Subscale scores range from 0 to 21, where a higher score represents a higher level of anxiety or depression.
Changes over the measurement points in the Infertility Questionnaire - Guilt/Blame subscale | Baseline, post-intervention: 4 weeks after the intervention initiation, 1-month follow-up, 5-year follow-up
  It has 5 items measuring participants' tendency to blame oneself or partner for infertility. Scores range from 5 to 25, where a higher score represent greater tendency to blame oneself or partner for infertility.
Changes over the measurement points in the 10-item Connor-Davidson Resilience Scale | Baseline, post-intervention: 4 weeks after the intervention initiation, 1-month follow-up, 5-year follow-up
  It has 10 items measuring participants' positive adaptation in the face of adversity. Scores range from 0 to 40, where a higher score represents a higher level of resilience.

OTHER OUTCOMES:
Satisfaction with Treatment Program Scale | Post-intervention: 4 weeks after the intervention initiation
  It has 5 items measuring participants' perceived satisfaction towards the couple-based I-BMS intervention for infertility. Only participants in the intervention group (arm 1) will complete it. Scores range from 5 to 25, where a high score represents greater satisfaction with the intervention.
Demographics | Enrolment: up to 8 weeks
  Single items will be used to gather information about participants' age, gender, education level, occupation, housing, monthly household income, and relationship status.
Infertility information: Cause of infertility | Enrolment: up to 8 weeks
  This will be retrieved from participants' medical records.
Infertility information: Year(s) of infertility | Enrolment: up to 8 weeks
  This will be retrieved from participants' medical records.
Infertility information: Previous assisted reproductive technology treatment | Enrolment: up to 8 weeks
  This will be retrieved from participants' medical records.
Infertility information: Previous reproductive history | Enrolment: up to 8 weeks
  This will be retrieved from participants' medical records.
Infertility information: Attitudes towards infertility | Enrolment: up to 8 weeks
  Four items are adopted from the Infertility Resilience Model assessment questionnaire. Participants will be asked: (a) who [they or their partner] feels more strongly about having children; (b) how long [in years] they are willing to keep trying to conceive; (c) the extent to which they understand how their partner feels about the infertility on a 5-point Likert scale ranging from 1 [never] to 5 [always]; and (d) the extent to which their partner understands how they feel about the infertility on a 5-point Likert scale ranging from 1 [never] to 5 [always]. Summative scores cannot be computed, but this outcome will be reported descriptively.
Marlow-Crowne Social Desirability Scale - Form C | Baseline
  It has 13 items measuring participants' tendency to present themselves in a favorable light. Scores range from 0 to 13, where a higher score represents a higher level of social desirability.
Cross-condition contamination check | Post-intervention: 4 weeks after the intervention initiation
  Two items will be used to control for the confounding effect of unexpected exposure to I-BMS intervention materials during the trial on primary outcomes. Only participants in the waitlist control group (arm 2) will complete it. Participants in the waitlist control group will be asked if they have: (a) viewed part or all of any I-BMS program materials; or (b) completed part or all of any I-BMS program homework/exercise. If they answer yes to any of these 2 items, they will be categorized as 1 [being exposed to I-BMS intervention materials]. If they answer no to these 2 items, they will be categorized as 0 [not being exposed to I-BMS intervention materials].
Medical outcomes | 5-year follow-up
  Participants' fertility treatment (e.g., types, recommendation) and outcomes (e.g., live birth, miscarriage) will be retrieved from their medical records.

CONTACTS AND LOCATIONS:
Overall Officials: Celia Hoi-Yan Chan, PhD, Principal Investigator — Department of Social Work and Social Administration, The University of Hong Kong
Locations (1):
- Department of Social Work and Social Administration, The University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No